CLINICAL TRIAL: NCT01475240
Title: A Cross-sectional Controlled Study to Evaluate the Impact of Hyperbilirubinemia on Markers of Cardiovascular Disease, Neurocognitive Function and Renal Markers in HIV-1 Infected Subjects on Protease Inhibitors
Brief Title: The Effect of Hyperbilirubinemia on CV Disease, Neurocog Function and Renal Function
Acronym: SSAT044
Status: Completed | Type: Observational
Sponsor: St Stephens Aids Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SSAT 044
Record Dates: First submitted 2011-10-31; First posted 2011-11-21 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: HIV
Keywords: HIV

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Controls: HIV-infected patients on stable > 6 months on TDF/FTC or ABC/3TC plus PI/r based ARV regimen with normal bilirubin
- Group 2: Cases: HIV-infected patients on stable >6 months on TDF/FTC or ABC/3TC plus PI/r based ARV regimen with HBR (>2.5 X upper limit)

SUMMARY:
Use of some protease inhibitors is associated with elevations of a blood pigment called bilirubin. This may occasionally lead to yellowing of the eyes (scleral icterus) or jaundice, but in the general population bilirubin elevations have been shown to have antioxidant and anti-inflammatory properties that could be associated with reduced risk of cardiovascular or other disease events.

Inflammation may also be relevant to neurocognitive impairment in HIV (Human Immunodeficiency Virus) infection hence elevations of bilirubin may also be protective against neurocognitive impairment.

The purpose of this study is to evaluate the impact of hyperbilirubinemia (HBR) on risk of heart and renal diseases, and cognitive function.

DETAILED DESCRIPTION:
Use of some protease inhibitors is associated with unconjugated hyperbilirubinemia as a result of inhibition of the UGT1A1 enzyme.

Elevated levels of unconjugated bilirubin are best characterized among individuals with Gilbert syndrome, which is the most common inherited cause of unconjugated hyperbilirubinemia, present in 3-10% of the general population. Gilbert syndrome arises through variants in the UGT1A1 enzyme, thus these PIs induce a biochemical picture similar to Gilbert syndrome. Although elevations of bilirubin may occasionally lead to scleral icterus or jaundice, cohort studies of individuals with Gilbert syndrome indicate bilirubin elevations may have antioxidant and anti-inflammatory properties and are associated with reduced risk of cardiovascular events.

Inflammation may also be relevant to cardiovascular (CV) risk, neurocognitive impairment and renal disease in HIV infection. This study seeks to investigate any association between antiretroviral associated HBR and CV risk markers, neurocognitive impairment and renal dysfunction

ELIGIBILITY:
Inclusion Criteria:

1. The ability to understand and sign a written informed consent form, prior to participation in any screening procedure and must be willing to comply with all study requirements.
2. Documented HIV-1 infection.
3. >18 years of age
4. Stable on PI based therapy with TDF/FTC or ABC/3TC > 6 months with either normal bilirubin or bilirubin >2.5 X upper limit
5. Stable for > 3 months on lipid lowering therapy, anticoagulant, hormone supplements, metformin (for lipohypertrophy) or other metabolic therapies
6. No known or past history of cardiovascular disease, neurocognitive disorder or renal disease.

Exclusion Criteria:

1. Grade 1-2 Bilirubin
2. Known CV disease (angina, coronary artery disease, peripheral vascular disease, stroke, congestive cardiac failure or myocardial dysfunction), Diabetes Mellitus, antihypertensive therapy
3. Chronic NSAID use including low dose aspirin
4. Known renal or CNS or neurocognitive disease
5. HIV RNA >400copies/ml in last 6 months
6. Change of antiretroviral Therapy in last 6 months
7. Active Hepatitis B (sAg +ve) or hepatitis C (detectable HCV RNA,, treated or cleared Hepatitis C permitted if infection and/or treatment > 6months previous)
8. Use of anabolic steroids. Cutaneous administered testosterone supplements stable for >3 months for documented hypogonadism permitted. Oral contraceptives stable for 3 months permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-infected males/females aged 18 years and above
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the impact of hyperbilirubinemia on markers of cardiovascular disease | 1 year
  Assessment of Pulse Wave Velocity; Carotid intimal thickness; Vascular markers (iCAM, vCAM); Lipid fractions and sub fractions

SECONDARY OUTCOMES:
To evaluate the impact of hyperbilirubinemia on neurocognitive function and renal markers | 1 year
  Assment of Neurocognitive testing; IL-6, d-dimer, uric acid, and hs-CRP; Urinary protein / creatinine ratio; Urinary Retinal binding / protein ratio

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Moyle, Dr, Principal Investigator — St Stephen's AIDS Trust
Locations (1):
- St Stephen's AIDS Trust, London, United Kingdom